CLINICAL TRIAL: NCT04473534
Title: Web Based Cognitive-behavioral Therapy in Patients With Obstructive Sleep Apnoea Syndrome and Insomnia: a Randomized Clinical Trial
Brief Title: Web Based CBT-I in Patients With OSA and Insomnia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely becauase of organisational problems.
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2361
Record Dates: First submitted 2020-07-10; First posted 2020-07-16 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea; Insomnia
Keywords: Obstructive sleep apnea; Insomnia; Web based CBT-I; CPAP treatment; Rehabilitation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm of CBT-I treatment (Experimental): Web cognitive behavioral therapy was administered before starting CPAP use by a psychologist expert in behavioral sleep medicine and expert in CBT-I. CBT-I was administered according to the same model and standard visual approach in patients with insomnia. Five sessions are scheduled: sleep psycho-education, sleep restriction, stimulus control, sleep hygiene and challenging beliefs and perception of sleep.
  Interventions: Behavioral: web based cognitive-behavioral therapy
- Arm of psycho-education session (Experimental): Single session of psycho-education about sleep, OSA, insomnia and interaction among them will be administered by web before beginning CPAP use
  Interventions: Behavioral: web based cognitive-behavioral therapy
- Arm of control TAU (Treatment As Usual) (No Intervention): The control group will receive TAU. Each patient will start to use CPAP after the diagnosis according to AASM (American Academy of Sleep Medicine) guideline.

INTERVENTIONS:
Behavioral: web based cognitive-behavioral therapy — one web session of psycho-education about sleep
  Other Names: Arm of psycho-education session
  Arms: Arm of CBT-I treatment; Arm of psycho-education session

SUMMARY:
Obstructive sleep apnea (OSA) and insomnia often occur in the same patient. Recent studies have demonstrated the efficacy of cognitive behavioral therapy (CBT-I) in patients with insomnia and OSA. Our aim is to verify the efficacy of web based CBT-I in patients with OSA and insomnia and the effect of web based CBT-I on the acceptance and adherence to CPAP (Continuous Positive Airway Pressure) therapy.

DETAILED DESCRIPTION:
Obstructive sleep apnea is one of the most common sleep disorders with high prevalence in males sex, is often associated with insomnia. The presence of both sleep disorders generates a vicious circle that exacerbates the clinical picture, makes difficult to accept and adhere to CPAP therapy and increase cardiovascular risk. CBT-I is considered the best treatment for insomnia and recent research has demonstrated the efficacy of CBT-I also when insomnia is associated with OSA. After six month of treatment we will test the efficacy of web-based CBT-I in patients with OSA and insomnia in comparison to one session of psycho education on sleep, OSA, insomnia, the interaction among them and the influence on CPAP adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Apnea-Hypopnea Index (AHI) ≥5

Exclusion Criteria:

* Complex sleep apnea
* AHI >35
* Psychiatric comorbidies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | Baseline
  Assessed by Insomnia Severity Index
Insomnia Severity | six months of CPAP use
  Assessed by Insomnia Severity Index

SECONDARY OUTCOMES:
Adherence to CPAP therapy | six months of use
  Hours of CPAP use during sleep with download of data

CONTACTS AND LOCATIONS:
Locations (1):
- Fabio Rossato, Veruno, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sweetman A, Lack L, Catcheside PG, Antic NA, Smith S, Chai-Coetzer CL, Douglas J, O'grady A, Dunn N, Robinson J, Paul D, Williamson P, McEvoy RD. Cognitive and behavioral therapy for insomnia increases the use of continuous positive airway pressure therapy in obstructive sleep apnea participants with comorbid insomnia: a randomized clinical trial. Sleep. 2019 Dec 24;42(12):zsz178. doi: 10.1093/sleep/zsz178. PMID 31403168
- [Background] Sweetman A, McEvoy RD, Smith S, Catcheside PG, Antic NA, Chai-Coetzer CL, Douglas J, O'Grady A, Dunn N, Robinson J, Paul D, Williamson P, Lack L. The effect of cognitive and behavioral therapy for insomnia on week-to-week changes in sleepiness and sleep parameters in patients with comorbid insomnia and sleep apnea: a randomized controlled trial. Sleep. 2020 Jul 13;43(7):zsaa002. doi: 10.1093/sleep/zsaa002. PMID 31927569